CLINICAL TRIAL: NCT03383887
Title: Effect of DAW1033D on Obstructive Sleep Apnea and Its Phenotypic Traits
Brief Title: DAW1033D in Obstructive Sleep Apnea
Acronym: OSAstimD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, David Andrew Wellman, Associate professor HMS, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014p001033D
Record Dates: First submitted 2017-12-13; First posted 2017-12-27 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo capsule 30 minutes before sleep
  Interventions: Drug: Placebo oral capsule
- DAW1033D (Active Comparator): DAW1033D capsule 30 minutes before sleep
  Interventions: Drug: DAW1033D oral capsule

INTERVENTIONS:
Drug: Placebo oral capsule — Placebo before sleep
  Arms: Placebo
Drug: DAW1033D oral capsule — DAW1033D before sleep
  Arms: DAW1033D

SUMMARY:
Obstructive sleep apnea (OSA) is common and has major health implications but treatment options are limited. OSA patients show a marked reduction in upper airway (UA) dilator muscle activity at sleep onset and this phenomenon leads to increased collapsibility of UA compared to normal subjects. In this protocol the investigators will test the effect of DAW1033D administered before sleep on OSA phenotype traits and OSA severity during sleep.

ELIGIBILITY:
Inclusion Criteria:

- AHI > 15

Exclusion Criteria:

* Any medical condition other than well controlled hypertension, diabetes, hyperlipidemia
* Any medication known to influence breathing, sleep/arousal or muscle physiology.
* Claustrophobia.
* Inability to sleep supine.
* Allergy to lidocaine, Oxymetazoline HCl, DAW1033D.
* Individuals with underlying cardiac disease, such as arrhythmias.
* Individuals taking psychiatric medications, or any of the studied medications for medical care.
* History of seizures
* For women: Pregnancy.
* History of panic disorder / hyperventilation syndrome / Attention deficit-hyperactivity disorder (ADHD) / autism

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep Disorders Research Program Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taranto-Montemurro L, Sands S, Azarbarzin A, Calianese N, Vena D, Hess L, Kim SW, White DP, Wellman A. Impact of cold and flu medication on obstructive sleep apnoea and its underlying traits: A pilot randomized controlled trial. Respirology. 2021 May;26(5):485-492. doi: 10.1111/resp.14009. Epub 2021 Jan 24. PMID 33491327

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo First, DAW1033D Second: Placebo-matching DAW1033D administered 30 mins before normal sleep time on first study night, then a 1-week non-treatment period, then DAW1033D administered 30 mins before normal sleep time on second study night.
- DAW1033D First, Placebo Second: DAW1033D administered 30 mins before normal sleep time on first study night, then a 1-week non-treatment period, then placebo administered 30 mins before normal sleep time on second study night.
Period: Overall Study
Arm/Group | Placebo First, DAW1033D Second | DAW1033D First, Placebo Second
Started | 5 | 6
Completed | 5 | 5
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Analyzed Participants: All participants who were randomized, completed both study nights, and were included in the analysis.
Arm/Group | All Analyzed Participants
Number analyzed (Participants) | 10
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [46 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Apnea Hypopnea Index (AHI, Events/Hour of Sleep)
Description: Based on previous studies the investigators anticipate that DAW1033D will reduce AHI more effectively in subjects with moderate sleep apnea, and mild to moderate pharyngeal collapsibility. AHI describes the frequency of obstruction of the upper airway during sleep and is commonly used to describe the presence and severity of obstructive sleep apnea.
Time Frame: 1 night
Population: 1 participant was not analyzed because he dropped out between the 2 intervention arms
Measure: Median (Inter-Quartile Range); unit: events/hour of sleep
Arm/Group | Placebo | DAW1033D
Number analyzed (Participants) | 10 | 10
events/hour of sleep | 21.6 [9.1 to 49.8] | 37.9 [5.1 to 55.4]
Statistical Analysis 1: Comparison: Placebo vs DAW1033D; Test type: Superiority; p = 0.56, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 2.7

2. Secondary Outcome: Collapsibility of the Upper Airway: VPassive
Description: Ventilation when ventilatory drive is relatively low during sleep
Time Frame: 1 night
Measure: Median (Inter-Quartile Range); unit: % eupneic ventilation
Arm/Group | Placebo | DAW1033D
Number analyzed (Participants) | 10 | 10
% eupneic ventilation | 74.8 [31.5 to 90.8] | 92.7 [70 to 97.2]
Statistical Analysis 1: Comparison: Placebo vs DAW1033D; Test type: Superiority; p = 0.027, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1 night
Arm/Group | Placebo | DAW1033D
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | DAW1033D (N=10)
insomnia (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-17): https://cdn.clinicaltrials.gov/large-docs/87/NCT03383887/Prot_SAP_000.pdf